CLINICAL TRIAL: NCT01622036
Title: The PreMiO Study: The Prevalence of Malnutrition in Oncology.
Brief Title: Prevalence of Malnutrition in Oncology (PreMiO)
Acronym: PreMiO
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Maurizio Muscaritoli, MD, Associated Professor, University of Roma La Sapienza
Other Study IDs: MM-SL-PreMIO
Record Dates: First submitted 2012-06-11; First posted 2012-06-18 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Malnutrition; Pre-cachexia; Cancer
Keywords: Malnutrition; pre-cachexia; cancer; cachexia; MNA; weight loss
MeSH Terms: conditions — Malnutrition; Neoplasms; Cachexia; Weight Loss

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer patients undergoing first medical oncology visit.

SUMMARY:
It is estimated that up to 30% of cancer patients die because of the effects of malnutrition, caused by a discrepancy between nutritional needs and intake (or utilization) of energy and essential nutrients. Malnutrition and its severe complication, cancer cachexia, are negative prognostic factors in neoplastic patients, inducing Decreased response and tolerance to antineoplastic treatments, decline in the functional status, reduced quality of life and reduced survival. Prevalence data on malnutrition in italian oncology patients are lacking and the available literature data on weight loss and malnutrition in oncology refer to patients in different phases of disease and therapy. Most importantly , strategies for prevention of malnutrition and cachexia in oncology are still largely disregarded and scarcely implemented.

The main objective of this project is to assess the prevalence of malnutrition in patients undergoing first medical oncology visit in Italy. Secondary objective is to increase awareness of metabolic and nutritional issues among medical oncologists, thus favoring the inclusion of metabolic-nutritional screening and monitoring in medical oncology protocols. This would in turn contribute to reduce the negative consequences of malnutrition- and cachexia-related complications.

DETAILED DESCRIPTION:
The acronym of the project "PreMiO" means "Prevalence of Malnutrition in Oncology".

The project arises from the observation that the negative consequences of cancer-related malnutrition and cachexia are still largely underestimated in most oncology units , both in Europe and the USA. Indeed, the prevention and treatment of the nutritional and metabolic sequelae of cancer and its treatment, are not perceived as a priority by most oncologists. This is quite surprising, considering the body of evidence demonstrating that the deterioration of the nutritional status adversely affects treatment response, morbidity, quality of life and survival of cancer patients. In other words, malnourished or cachectic cancer patients lose chances to be adequately treated for their underlying disease. Approximately one quarter of all deaths in western society are due to cancer. Half of all patients with cancer lose body weight; one third lose more than 5% of their original body weight and up to 20% of all cancer deaths are caused directly by cachexia. The greatest prevalence of weight loss is seen among patients with solid tumours: gastric, pancreatic, lung, colorectal, and head and neck. The overall prevalence of weight loss in cancer patients may rise as high as 86% in the last 1-2 weeks of life.The pathogenesis of weight loss, malnutrition and cachexia in cancer is multifactorial and represent the result of the complex interplay between the tumor, host's metabolism, tumor-derived and host-derived humoral factors, and the negative consequences of anticancer treatments on the patient's ability to assume, absorb and metabolize nutrients.

Objectives The objective of the PreMiO project is to obtain data on the prevalence of malnutrition in Italian cancer patients undergoing the first medical oncology visit. The project is innovative since an oncologist, not a nutrition specialist, will perform the nutritional evaluation of the patients.

The data obtained will contribute to increase the awareness of metabolic and nutritional problems in oncology, favoring the inclusion of the initial assessment and nutritional-metabolic monitoring in oncological protocols.

Patients and Methods "PreMIO" will be a prospective, multicentre observational study, designed to assess the nutritional status in cancer patients presenting for the first visit to an oncological center. Enrollment will be conducted at Italian ESMO-accredited centers and in other medical oncological centers in Italy. Six-thousand patients have been considered an adequate sample for a suitable estimation of the prevalence of malnutrition in Italian cancer patients at first medical oncology visit. Patient recruitment will be ensured through enrollment by 60 centers throughout the Italian national territory (North, Center, South). The instruments used for patients' evaluation will be the Mini Nutritional Assessment ® (MNA ®) and the criteria for the diagnosis of pre-cachexia elaborated by ESPEN. Pre-cachexia is a clinical condition characterized , in the context of a chronic disease (i.e. cancer), by unintentional weigh loss ≤ 5% during last 6 months, chronic systemic inflammation and anorexia or anorexia-related symptoms. Although other nutritional tools are available for nutritional status evaluation (Nutritional Risk Screening 2002, NRS 2002; Malnutrition Universal Screening Tool, MUST), even in oncological setting (Subjective Global Assessment, SGA; Patient-Generated Subjective Global Assessment, PG-SGA), we choose MNA® for its diagnostic sensitivity and its rapidity of administration. The MNA ® consists of a first screening part and of a second part as global assessment, which allows to obtain a score reflecting the patient nutritional status. Moreover, this instrument was recently considered the best screening method of nutrition status in patients with metastatic lung cancer. The data generated in each participating center will be collected by the Coordinator Centre (IDI-IRCCS). Patients will be stratified according to cancer type and localization, disease stage, age, sex, general condition. It is expected that the prevalence of malnutrition and pre- cachexia will vary widely, depending on tumor type, localization, stage and previous surgical treatment. Multivariate analysis will allow to discriminate among the factors contributing to the occurrence and prevalence of malnutrition in the study population.

ELIGIBILITY:
Inclusion Criteria:

* patients at first medical oncology visit
* diagnosis of solid tumor
* age > 18 years
* no previous anticancer therapies (e.g. radiotherapy or chemotherapy)
* Life expectancy >3 months according with PaP score
* Informed consent

Exclusion Criteria:

* Oral feeding incapacity or intestinal obstruction
* Decompensated metabolic disorders
* Severe liver failure (total bilirubin >1.5 mg/dL (25μmol/L), and AST (SGOT)/ ALT (SGPT) >2 x ULN or, in the case of metastatic liver, > 5 x ULN) or severe kidney failure (creatinine > 2.0 mg/dL (177 μmol/L), creatinine clearance ClCr < 50ml/min).
* Acute Decompensated heart failure
* Active infection
* Primary brain tumors or metastatic brain tumors
* severe psychiatric disorders
* MMSE < 25/30 (in patient aged >70).
* Inadequate logistical support for the study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment will be conducted at Italian ESMO-accredited centers and in other medical oncological centers in Italy. Six-thousand patients have been considered an adequate sample for a suitable estimation of the prevalence of malnutrition in Italian cancer patients at first medical oncology visit. Patient recruitment will be ensured through enrollment by 60 centers throughout the Italian national territory (North, Center, South and Islands).
Sampling Method: Probability Sample
Enrollment: 1978 (Actual)
Dates: Start 2012-06; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Malnutrition | Assessed at the first medical oncology visit
  Malnutrition will be assessed by Mini Nutritional Assessment, biochemical analysis and diagnostic criteria of pre-cachexia.

SECONDARY OUTCOMES:
Anorexia | Assessed at the first medical oncology visit
  Anorexia will be assessed via a modified version of AC/S-12 FAACT, via Visual Analogue Scale and specific questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Rome, Italy

REFERENCES:
- [Result] Muscaritoli M, Bossola M, Aversa Z, Bellantone R, Rossi Fanelli F. Prevention and treatment of cancer cachexia: new insights into an old problem. Eur J Cancer. 2006 Jan;42(1):31-41. doi: 10.1016/j.ejca.2005.07.026. Epub 2005 Nov 28. PMID 16314085
- [Result] Laviano A, Meguid MM, Rossi-Fanelli F. Cancer anorexia: clinical implications, pathogenesis, and therapeutic strategies. Lancet Oncol. 2003 Nov;4(11):686-94. doi: 10.1016/s1470-2045(03)01247-6. PMID 14602249
- [Result] Tisdale MJ. Mechanisms of cancer cachexia. Physiol Rev. 2009 Apr;89(2):381-410. doi: 10.1152/physrev.00016.2008. PMID 19342610
- [Result] Dewys WD, Begg C, Lavin PT, Band PR, Bennett JM, Bertino JR, Cohen MH, Douglass HO Jr, Engstrom PF, Ezdinli EZ, Horton J, Johnson GJ, Moertel CG, Oken MM, Perlia C, Rosenbaum C, Silverstein MN, Skeel RT, Sponzo RW, Tormey DC. Prognostic effect of weight loss prior to chemotherapy in cancer patients. Eastern Cooperative Oncology Group. Am J Med. 1980 Oct;69(4):491-7. doi: 10.1016/s0149-2918(05)80001-3. PMID 7424938
- [Result] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Result] Muscaritoli M, Anker SD, Argiles J, Aversa Z, Bauer JM, Biolo G, Boirie Y, Bosaeus I, Cederholm T, Costelli P, Fearon KC, Laviano A, Maggio M, Rossi Fanelli F, Schneider SM, Schols A, Sieber CC. Consensus definition of sarcopenia, cachexia and pre-cachexia: joint document elaborated by Special Interest Groups (SIG) "cachexia-anorexia in chronic wasting diseases" and "nutrition in geriatrics". Clin Nutr. 2010 Apr;29(2):154-9. doi: 10.1016/j.clnu.2009.12.004. Epub 2010 Jan 8. PMID 20060626
- [Result] Lennard-Jones JE, Arrowsmith H, Davison C, Denham AF, Micklewright A. Screening by nurses and junior doctors to detect malnutrition when patients are first assessed in hospital. Clin Nutr. 1995 Dec;14(6):336-40. doi: 10.1016/s0261-5614(95)80050-6. PMID 16843954
- [Result] Muscaritoli M, Molfino A, Lucia S, Rossi Fanelli F. Cachexia: a preventable comorbidity of cancer. A T.A.R.G.E.T. approach. Crit Rev Oncol Hematol. 2015 May;94(2):251-9. doi: 10.1016/j.critrevonc.2014.10.014. Epub 2014 Nov 7. PMID 25468676
- [Result] Muscaritoli M, Aversa Z, Lucia S. The conundrum of pre-cachexia existence. Clin Nutr. 2014 Dec;33(6):1160. doi: 10.1016/j.clnu.2014.09.024. No abstract available. PMID 25453398
- [Result] Lucia S, Esposito M, Rossi Fanelli F, Muscaritoli M. Cancer cachexia: from molecular mechanisms to patient's care. Crit Rev Oncog. 2012;17(3):315-21. doi: 10.1615/critrevoncog.v17.i3.90. PMID 22831162
- [Result] Gioulbasanis I, Baracos VE, Giannousi Z, Xyrafas A, Martin L, Georgoulias V, Mavroudis D. Baseline nutritional evaluation in metastatic lung cancer patients: Mini Nutritional Assessment versus weight loss history. Ann Oncol. 2011 Apr;22(4):835-841. doi: 10.1093/annonc/mdq440. Epub 2010 Oct 11. PMID 20937647